CLINICAL TRIAL: NCT05137782
Title: The Science of the Art of Palliative Care Pilot
Brief Title: The Science of the Art of Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Amber Barnato, Director, The Dartmouth Institute, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02001223
Record Dates: First submitted 2021-11-17; First posted 2021-11-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Gastrointestinal Cancer; Lung Cancer; Advanced Cancer
Keywords: Palliative Care
MeSH Terms: conditions — Gastrointestinal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Patients and care partners receive specialty primary care and participate in pre- and post- functional MRI scans to measure the effects of the specialty palliative care intervention.
  Interventions: Other: Specialty Palliative Care

INTERVENTIONS:
Other: Specialty Palliative Care — Specialty palliative care, as opposed to primary palliative care.

SUMMARY:
This feasibility pilot study is designed to learn whether patients and their care partners (e.g., family members) are willing and able to complete two study visits at Dartmouth College while receiving cancer care at Dartmouth-Hitchcock Medical Center.

DETAILED DESCRIPTION:
A feasibility pilot open label, single-arm observational case series of 10 patients with metastatic gastrointestinal and lung cancer patients and 10 care partners. Participants will complete two study visits, separated by approximately 8-16 weeks of usual oncologic care with early integrated specialty palliative care. The palliative care physician will also be a study participant.

Primary Objective: To develop and refine study procedures which can be used in future research in order to further understanding of the mechanisms of action of specialty palliative. Expected products: manual of operating procedures and web-based data collection forms.

Secondary Objectives: To test the feasibility of conducting a mechanism-focused clinical trial of primary palliative care vs. specialty palliative care for advanced cancer patients and their care partners. Expected products: preliminary data demonstrating the feasibility of study procedures sufficient to prove this study design is possible.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patient: has received a diagnosis of advanced lung or gastrointestinal cancer within the last 24 weeks (note: advanced GI cancer will likely be pancreatic or colorectal)
* Care partner: care partner of a patient who has received a diagnosis of metastatic lung or gastrointestinal cancer who has provided consent for study (either with our without functional MRI study visits)
* Be able to understand study requirements and make an informed decision to participate
* Be able to speak and read English

Exclusion Criteria:

* Life expectancy of <8 weeks
* Known brain metastases
* Claustrophobia
* Both patient and care partner refuse to participate in fMRI scan (ie., either patient or care partner must agree to an fMRI scan in order for either to participate)
* Contraindications to MRI (e.g.: implanted or embedded metal/metal fragments. Metals in the body make the participant unable to undergo an MRI which makes them ineligible for study participation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Operationalization as measured by the creation of a manual of operating procedures and web-based data collection forms | 6 months
  Establish acceptable operating procedures and data collection instruments which can be replicated for future projects.

SECONDARY OUTCOMES:
Feasibility as measured by participant interest | 6 months
  Percent of participants approached and interested in participating
Feasibility as measured by enrollment number | 6 months
  Percent of participants approached and enrolled
Feasibility as measured by willingness to be randomized | 6 months
  Percent of participants enrolled and willing to be randomized
Feasibility as measured by procedure completion rate | 6 months
  Percent of participants randomized and completed procedures (specialty palliative care, fMRIs, surveys, bio response measurements).
Feasibility as measured by participant withdrawal rate | 6 months
  Percent of participants not completing each study visit and specialty primary care visit
Tolerability as measured by subjective units of distress scores (SUDS, 0-100) | 6 months
  The SUDs Rating Scale, or Subjective Units of Distress Scale (SUDs) as it is officially known, is used to measure the intensity of distress or nervousness in people with social anxiety. The SUDs is a self-assessment tool rated on a scale from 0 to 100.
Tolerability as measured by rates of study procedure non-completion. | 6 months
  Percent of participants not completing each study procedures (specialty palliative care, fMRIs, surveys, bio response measurements).
Acceptability as measured by response to questions of level of burden. | 6 months
  Two closed-ended Likert scale items regarding study burdensomeness. (this investigator-created instrument is in development)
Acceptability as measured by willingness to recommend study participation to others. | 6 months
  Measured by the Net Promoter Score - The Net Promoter Score is an index that measures the willingness of participants to recommend a services to others. It is used as a proxy for gauging overall satisfaction with a service. Net Promoter Score (scale from 0 to 10 with 3 groups: promoters for 9-10, passive for 7-8 and detractor for below 6).

CONTACTS AND LOCATIONS:
Overall Officials: Amber Barnato, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No